CLINICAL TRIAL: NCT06768476
Title: Phase I Trial of CART123 Cells Given in Combination With Ruxolitinib in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: CART123 + Ruxolitinib in Relapsed/Refractory AML
Acronym: AML
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 50424
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed AML; Refractory AML
Keywords: CART; refractory; relapsed; acute; myeloid; leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: DL1 (Experimental): * LD Chemo: Day -6 to Day -4 (±1d)
  * Ruxolitinib: Daily beginning on Day -6 (±1d) through D14 post CART123 infusion.
  * CART123 Cells: Single infusion on Day 0
  Interventions: Biological: CART123 Cells; Drug: Ruxolitinib 10 MG
- Arm A: DL-1 (Experimental): * LD Chemo: Day -6 to Day -4 (±1d)
  * Ruxolitinib: Daily beginning on Day -6 (±1d) through D14 post CART123 infusion.
  * CART123 Cells: Single infusion on Day 0
  Interventions: Biological: CART123 Cells; Drug: Ruxolitinib 5 MG
- Arm B: DL-1 (Experimental): * LD Chemo: Day -6 (-1d) to Day -2 (-1d)
  * Venetoclax: Day -6 (-1d) through Day +7 - Day +14 post-CART123 infusion
  * Ruxolitinib: Daily beginning on Day -1 through Day +7 post CART123 infusion.
  * CART123 Cells: Single infusion on Day 0
  Interventions: Biological: CART123 Cells; Drug: Ruxolitinib 5 MG

INTERVENTIONS:
Biological: CART123 Cells — 1.3x10^8 CART123 cells
Drug: Ruxolitinib 10 MG — Twice Daily
  Arms: Arm A: DL1
Drug: Ruxolitinib 5 MG — Twice Daily
  Arms: Arm A: DL-1; Arm B: DL-1

SUMMARY:
Phase I, open-label study to assess the safety, feasibility, pharmacokinetics, and preliminary efficacy of CART123 cells given in combination with ruxolitinib in patients with relapsed or refractory acute myeloid leukemia (AML). All subjects will receive a single infusion of CART123 cells following ruxolitinib administration and lymphodepletion. Ruxolitinib dosing will begin at initiation of lymphodepleting chemotherapy (Day -6 ±1d) and continue for up to 14 days post CART123 administration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed informed consent form 2. Male or female age ≥ 18 years. 3. Patients with active acute myeloid leukemia (AML) with no available curative treatment options using currently available therapies. This is specifically defined as one of the following:

  1. AML that has not achieved a complete remission or morphologic leukemia free state by ELN 2022 criteria57 after at least 2 cycles of induction (includes partial remission or refractory/primary refractory disease), OR:
  2. AML relapsed following allogeneic stem cell transplantation (including MDS evolved to AML post-allogeneic stem cell transplant).

  i. Note: Morphologic relapse is not required; Patient may have persistent/recurrent disease-associated molecular, phenotypic or cytogenetic abnormalities (i.e., MRD) at any time after allogeneic HCT to qualify. Mutations involving DNMT3A, ASXL1 or TET2 should not count as molecular MRD+ disease unless accompanied by other, more specific disease-related molecular or cytogenetic abnormalities.

  4. Patients with relapsed disease after prior allogeneic SCT must be at least 3 months from transplantation (where receipt of the stem cell product is defined as day 0) and must not require systemic immunosuppression (for prevention or treatment of GVHD).

  5. Patients must have a suitable stem cell donor identified with projected ability to proceed to transplant within 6-8 weeks of CART123 infusion if clinically indicated. Donor may be matched or mismatched and must be found to be suitable according to the institution's standard criteria.

  6. Adequate organ function defined as:
  1. Estimated creatinine clearance > 35mL/min using the CKD-EPI equation for Glomerular Filtration Rate (GFR); Patients must not be on dialysis
  2. ALT/AST ≤ 5x upper limit of normal range
  3. Direct bilirubin ≤ 2.0 mg/dl, unless the subject has Gilbert's syndrome (≤3.0 mg/dl)
  4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
  5. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by transthoracic echocardiography or MUGA scan.

     7. ECOG Performance Status 0-2.

     Exclusion Criteria:
* 1. Patients with the JAK2 V617F mutation by PCR or next generation sequencing. 2. Patients with signs or symptoms indicative of active CNS involvement. A CNS evaluation should be performed as clinically appropriate to rule out CNS involvement.

  3. Patients with relapsed AML with t(15:17). 4. Active hepatitis B, active hepatitis C, or other active, uncontrolled infection.

  5. Active acute or chronic GVHD requiring systemic therapy. 6. Class III/IV cardiovascular disability according to the New York Heart Association Classification.

  7. Clinically apparent arrhythmia or arrhythmias that are not stable on medical management within two weeks of physician-investigator confirmation of eligibility.

  8. Dependence on systemic steroids or immunosuppressant medications. For additional details regarding use of steroid and immunosuppressant medications.

  9. Planned use of fluconazole within the anticipated study treatment window. For additional details on concomitant medication restrictions.

  10. Receipt of prior CART123 therapy. 11. Pregnant or nursing (lactating) patients. Participants of reproductive potential must agree to use acceptable birth control methods.

  12. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.

  13. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2045-03 (Estimated); Study Completion 2045-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of CART123 cells when given in combination with ruxolitinib | 15 Years
  Type, frequency, severity, and attribution of AEs/SAEs, including the incidence and severity of IEC-associated adverse events.
Evaluate the safety of CART123 cells when given in combination with ruxolitinib | 3 months
  Occurrence of treatment-limiting toxicities (TLTs)
Evaluate the safety of CART123 cells when given in combination with ruxolitinib | 3 months
  The proportion of subjects requiring ruxolitinib dose modifications by assigned dose.

SECONDARY OUTCOMES:
Evaluate study feasibility | 3 months
  The proportion of eligible subjects who receive both investigational products as per protocol.
Evaluate study feasibility | 3 months
  The proportion of eligible subjects who receive all planned doses of ruxolitinib.
Describe preliminary efficacy of CART123 cells given in combination with ruxolitinib | From enrollment to Day 28, post treatment.
  Objective Response Rate (ORR) at Day 28
Describe preliminary efficacy of CART123 cells given in combination with ruxolitinib | 15 years
  Duration of Response (DOR)
Describe preliminary efficacy of CART123 cells given in combination with ruxolitinib | 15 Years
  Progression-free survival (PFS)
Describe preliminary efficacy of CART123 cells given in combination with ruxolitinib | 15 Years
  Overall Survival (OS)
Describe preliminary efficacy of CART123 cells given in combination with ruxolitinib | From enrollment to Day 28, post treatment.
  Reduction of blast count in the peripheral blood and marrow using standard clinical criteria (CBC with differential count, marrow aspirate with differential count) and flow cytometry at Day 28
Describe preliminary efficacy of CART123 cells given in combination with ruxolitinib | 15 Years
  Percentage of subjects undergoing alloHCT

CONTACTS AND LOCATIONS:
Overall Officials: Saar Gill, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No